CLINICAL TRIAL: NCT04377971
Title: The Effectiveness of the Teach-back Method on Patient Satisfaction and Adherence to Wound Care Regimen After Mohs Micrographic Surgery: A Pilot Study
Brief Title: Teach-back Method on Patient Satisfaction and Adherence to Wound Care Regimen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CASE1620
Record Dates: First submitted 2020-05-04; First posted 2020-05-07 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Keratinocyte Carcinoma
Keywords: Mohs Micrographic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ask-tell-ask method (Experimental): Study team will provide participant education using the ask-tell-ask method. Participants will receive a post-operative instruction sheet containing detailed information regarding wound care for reference and will receive a phone call at 1 week to inquire about wound care adherence. Participants will come to clinic at 2 weeks to have wounds assessed in addition to answering surveys regarding wound care adherence and participant experience.
  Interventions: Behavioral: Ask-tell-ask education; Other: Participant satisfaction survey; Other: Wound care adherence survey
- Standard of Care (SOC) (Active Comparator): Participants will receive SOC education from the researcher. Participants will receive a post-operative instruction sheet containing detailed information regarding wound care for reference and will receive a phone call at 1 week to inquire about wound care adherence. Participants will come to clinic at 2 weeks to have wounds assessed in addition to answering surveys regarding wound care adherence and participant experience.
  Interventions: Behavioral: SOC education; Other: Participant satisfaction survey; Other: Wound care adherence survey

INTERVENTIONS:
Behavioral: SOC education — Standard participant education from researcher
  Arms: Standard of Care (SOC)
Behavioral: Ask-tell-ask education — Participant education using the ask-tell-ask method. First the researcher will ask a question about participant understanding of wound care and after hearing the participant's answer, the researcher will then proceed to tell the patient how to best take care of their wound using a standardized script. After the educational portion, the researcher will then ask the patient to repeat the information that was shared. If the participant's answer is wrong or incomplete, the researcher will then explain the instructions again to ensure that the participant understands the steps needed.
  Arms: Ask-tell-ask method
Other: Participant satisfaction survey — Participant satisfaction survey using components of the 16 item Skindex questionnaire and the 18 item version Patient Satisfaction Survey, adapted for treatment of skin cancer to characterize patient experience administered at two weeks post-operatively in person
Other: Wound care adherence survey — Wound care adherence survey administered at one week over the phone and at two weeks in person

SUMMARY:
The purpose of this study is to examine a different way to educate patients about taking care of their wound and see how this method affects patient satisfaction, compliance to the wound care regimen, and patient experience.

The teach-back method is delivered using the ask-tell-ask method. Investigators will ask the patient about their knowledge of wound care healing, provide the patient educational component, then ask the patient to repeat what was said. If the answer is wrong or incomplete, the researcher will go over the information again with the patient to clear up any misunderstandings.

DETAILED DESCRIPTION:
Patients undergoing Mohs Micrographic surgery for skin cancers on the lower extremities for the first time that are left to heal by secondary intention are randomized either to receive a scripted teach-back session or a standard of care wound care education. This study wishes to compare wound care adherence, patient experience, wound complications, and the number of phone calls made by patients to the office between the two cohorts

primary objective is to determine whether study participants who have received the teach-back method have an increase wound care adherence at one week post-operatively, compared to those who received the standard of care.

To characterize differences in the patient experience between the two interventional groups 2 weeks after surgery.

To determine whether the number of phone calls made post-operatively by patients will decrease in a 2 week follow-up time period.

To characterize the differences in patient wound care adherence at 2 weeks after surgery.

To determine whether there is a difference in complication incidence post-operatively

ELIGIBILITY:
Inclusion Criteria:

* Presenting to outpatient Mohs clinic at University Department of Dermatology, Two Chagrin Highlands for the first time
* Have excision(s) from Mohs Micrographic Surgery on the lower extremities that are left to heal by secondary intention
* English-speaking

Exclusion Criteria:

* Non-English speaking
* A clinical diagnosis of mental, learning, and visual disabilities
* A clinical diagnosis of dementia
* Those who have received Mohs Micrographic Surgery before regardless of area

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Wound care adherence as measured by wound care adherence survey | 1 week
  Wound care adherence as measured by a wound care adherence survey with scale values ranging from 3-15, with a higher score indicating greater compliance
  Independent two-sample two-sided t-tests to compare wound care adherence scores between the intervention group (receiving the "teach-back method") and the control group (receiving the standard of care).

SECONDARY OUTCOMES:
Patient experience as measured by participant satisfaction survey | At 2 weeks
  Patient experience as measured by participant satisfaction survey, which uses components of the 16 item Skindex questionnaire and the 18 item version Patient Satisfaction Survey, adapted for treatment of skin cancer to characterize patient experience. The survey scale ranges from 4-20, with a higher score indicating a greater patient experience.
Number of phone calls made post-operatively by participants | At 2 weeks
  Number of phone calls made post-operatively by participants
Complication incidence post-operatively | At 2 weeks
  Complication incidence post-operatively
Wound care adherence as measured by wound care adherence survey | At 2 weeks
  Wound care adherence as measured by a wound care adherence survey with scale values ranging from 3-15, with higher scores indicating greater compliance.
  Independent two-sample two-sided t-tests to compare wound care adherence scores between the intervention group (receiving the "teach-back method") and the control group (receiving the standard of care)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Wong, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
We will not share IPD in order to protect the identity of the research participants